CLINICAL TRIAL: NCT03022448
Title: Geriatric Assessmen of Elderly "Unsuited" Patients Receiving Trabectedin in First Line Treatment For Advanced Soft Tissue Sarcomas (STS)
Acronym: E-TRAB
Status: Completed | Type: Observational
Sponsor: GWT-TUD GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: E-Trab
Record Dates: First submitted 2017-01-13; First posted 2017-01-16 (Estimated); Last update posted 2022-04-04 (Actual); Status verified 2022-04

CONDITIONS: Advanced Soft-tissue Sarcoma; Metastatic Soft-tissue Sarcoma
Keywords: soft tissue sarcomas (STS); trabectedin; metastatic STS patients; overall survival
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treatment Group: Trabectedin will be used according to the local SmPC. Modification of the treatment schedule should follow the standard medical practice at the discretion of the treating physician and is not part of this Observational Plan.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a NIS. No intervention.

SUMMARY:
The aim of the non-interventional study is to prospectively collect and analyze data on the geriatric assessment of patients undergoing systemic 1st line therapy with trabectedin with focus on patients who have been assessed by the treating physician as being unsuited to receive standard chemotherapy with anthracyclines and / or ifosfamide.

Trabectedin will be used according to the local SmPC. Modification of the treatment schedule should follow the standard medical practice at the discretion of the treating physician and is not part of this Observational Plan.

ELIGIBILITY:
Inclusion Criteria:

Written informed consent

* Age of ≥ 60 years at study inclusion with a limited number of "unsuited" patients younger than 60 years
* Histologically proven advanced and/or metastatic STS, intermediate/high grade
* Presence of measurable disease according to RECIST 1.1. (optional, according to local clinical practice)
* Patients indicated for 1st line treatment with trabectedin according to local SmPC
* ECOG Performance Status 0, 1 or 2
* bone marrow function according to local SmPC
* hepatic function according to local SmPC
* Ability to understand and follow study-related instructions

Exclusion Criteria:

* Histologically proven advanced and/or metastatic STS of the following tumor types:
* Embryonal rhabdomyosarcoma
* Chondrosarcoma (excluding extraskeletal myxoid chondrosarcoma)
* Osteosarcoma (excluding extraskeletal osteosarcoma)
* Ewing tumors/primitive neuroectodermal tumor
* Gastrointestinal stromal tumors
* Dermatofibrosarcoma protuberans
* Use of any investigational agent within 28 days prior to treatment start
* Exclusion periods from other studies or simultaneous participation in other clinical studies
* Contraindications according to the local SmPC of Yondelis® (see Appendix A)
* Subject is in custody by order of an authority or a court of law
* Previous assignment to the E-Trab study (An individual subject may only be included once in the study)
* Criteria which in the opinion of the investigator preclude participation for scientific reasons, for reasons of compliance, or for reasons of the subject's safety

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elderly patients with advanced and/or metastatic STS (≥ 60 years including a maximum of 1/6 of "unsuited" patients younger than 60 years)
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | 12 month after LPFV
  Overall survival for each patient will be followed until the end of the study that is defined by 12 months after inclusion of the last patient.

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Kasper, Prof., Principal Investigator — University of Heidelberg Mannheim University Medical Center Interdisciplinary Tumor Center, Sarcoma Unit
Locations (12):
- Austria (2):
  - Klinikum Klagenfurt am Wörthersee, Klagenfurt
  - Medizinische Universität Wien, Vienna
- Germany (8):
  - HELIOS Klinikum Bad Saarow, Bad Saarow
  - HELIOS Klinikum Berlin Buch, Berlin
  - Klinikum Spandau, Berlin
  - Universitätsklinikum Carl Gustav Carus der TU Dresden, Dresden
  - Universitätsklinikum Heidelberg, Heidelberg
  - University of Heidelberg Mannheim University Medical Center Interdisciplinary Tumor Center, Sarcoma Unit, Mannheim
  - Klinikum Nürnberg Nord, Nuremberg
  - Universitätsklinikum Ulm, Ulm
- Switzerland (2):
  - Universitätsspital Bern, Bern
  - Kantonsspital St. Gallen, Sankt Gallen

IPD SHARING:
Plan to Share IPD: No